CLINICAL TRIAL: NCT01403727
Title: Electromagnetic Tracking of Devices During Biopsy Procedures
Status: Completed | Type: Observational
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 2010_MtSinai_BiopTrial_V2
Record Dates: First submitted 2011-07-22; First posted 2011-07-27 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Liver Tumors
Keywords: Biopsy of liver tumors
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Unassisted Biopsy - CONTROL GROUP: Routine biopsy needle placement and Physician blinded to needle location
- Assisted Biopsy - STUDY GROUP: The physician will be shown the PercuNav screen and will correct the desired approach path.

SUMMARY:
The purpose of the trial is to evaluate the differences between PercuNav assisted and unassisted biopsy in the areas of CT radiation dose, procedure time and biopsy accuracy.

This prospective, randomized, controlled trial will compare the use of electromagnetic tracking and image guidance (CT) during biopsy procedures verses the typical CT image guided procedure alone.

DETAILED DESCRIPTION:
The purpose of the trial is to evaluate the differences between PercuNav assisted and unassisted biopsy. The primary objective of this study is to assess and quantify any differences between assisted and unassisted CT guided biopsy procedures of the liver with respect to radiation dose.

The secondary objectives of this study are to assess and quantify any differences between assisted and unassisted CT guided biopsy procedures with respect to:

* Total procedure time
* Accuracy of needle targeting (distance from defined target on PercuNav and angle of entry)
* Number of needle passes
* Target registration error (TRE- distance between "virtual" needle position (tracking data) and the actual needle position (CT confirmation scan))

The study will consist of 50 patients from 1 site. The expected completion time for enrollment is 3 months, but will depend on the ability of the clinic to enroll patients. There are two arms in the study. An Unassisted Biopsy Control arm (physician and patient blinded to needle positioning using PercuNav system) and Assisted Biopsy (Physician not blinded to needle positioning using PercuNav). Patients will be randomized to each arm.

The PercuNav provides real-time, three-dimensional visualization and navigation tools for all stages of diagnosis and surgery including pre-procedure planning and intra-procedure navigation. PercuNav transforms two-dimensional patient images (scan sets), derived from CT, PET/CT and MRI into dynamic representations on which a tool can be navigated and fused with ultrasound. The system performs spatial mapping from one image space to another image space or from image space to physical space (registration) allowing the physician to correlate scan sets with each other and to the patient.

For this trial, each patient will have a pre-procedure CT image set of the area of interest. The image set should display the patient in the same position that the biopsy will be performed in, although not requisite.

Unassisted Biopsy - CONTROL GROUP (Physician blinded to PercuNav system):

The tracking device will be placed on the patient's skin at the desired point of entry. Without displaying the PercuNav screen to the physician, a screen capture will be taken to record the approach path. At the point of insertion, the time stamp will be recorded and the start button will be pressed. Once the physician states they are at the defined target a screen capture will be taken on the PercuNav and the distance to target and time stamp will be recorded by pushing the start button again.

The final dose of radiation displayed by the CT scanner will be recorded on the Case Report Form.

Assisted Biopsy - STUDY GROUP:

The tracking device will be placed on the patient's skin at the desired point of entry. Without displaying the PercuNav screen to the physician, a screen capture will be taken to record the approach path. The physician will be shown the PercuNav screen and will correct the desired approach path and another screen capture will be taken. At the point of insertion, the time stamp will be recorded and the start button will be pressed. Once the physician states they are at the defined target a screen capture will be taken on the PercuNav and the distance to target and time stamp will be recorded.

The final dose of radiation displayed by the CT scanner will be recorded on the Case Report Form.

The primary study objective is to quantify, in terms of a point estimate and confidence interval, the treatment effect which characterizes the mean difference in number of CT scans between the "unassisted" CT and "assisted" CT groups during guided liver biopsy procedures. More specifically, the goal will be to show with 95% Confidence that the "assisted" CT procedure leads to 3 fewer scans, on average, than the "unassisted" CT group during guided liver biopsies.

H0: uT - aT < 3 scans HA: uT - aT >= 3 scans uT = mean number of scans during "unassisted" CT procedure aT = mean number of scans during "assisted" CT procedure Equivalently, the desired superiority will have been demonstrated whenever the lower 95% confidence limit on the difference, "unassisted" CT minus "assisted" CT, exceeds 3 scans.

Primary Endpoint and Objective:

The primary endpoint for this study is the number of CT radiation exposure scans received during the course of a CT guided liver biopsy procedure. The primary study objective is to characterize the difference in the number of scans received between the "assisted" and the "unassisted" CT groups during guided liver biopsy procedures.

The primary measure that will be assessed and quantified is any differences between assisted and unassisted CT guided liver biopsies with respect to radiation dose.

The secondary measures that will be assessed and quantified are any differences between assisted and unassisted CT guided procedures with respect to:

* Total procedure time
* Accuracy of needle targeting (distance from defined target on PercuNav and angle of entry)

ELIGIBILITY:
Inclusion Criteria:

1. Has had a pre-operative CT scan performed and will be undergoing a biopsy procedure of the liver;
2. Is over the age of 18;
3. Has the ability to understand and the willingness to sign a written informed consent form, and complies with the protocol;
4. Has the ability to follow procedural instructions, including, but not limited to, holding their breath and remaining reasonably motionless during the procedure.

Exclusion Criteria:

1. Was precluded from a biopsy procedure based on standard exclusions;
2. Has an adhesive allergy (due to the application of active fiducials with adhesive backing);
3. Has a pacemaker or automatic implantable cardiac defibrillator;
4. Has a gross body weight above 180lbs for women and 260lbs for men;
5. Is pregnant

A patient may be excluded after enrollment if any of the following criteria are met:

1. The patient's health and/or safety become jeopardized for any reason making it unsafe to continue; 2. Technical errors and/or difficulties; 3. Any reasonable rationale put forth by the physician or investigator 4. Lost to follow up - In-evaluable data

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a liver biopsy procedure
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Radiation Dose | 24 hrs
  The primary objective of this study is to assess and quantify any differences between assisted and unassisted CT guided biopsy procedures of the liver with respect to radiation dose.

SECONDARY OUTCOMES:
Total procedure time | 24 hrs
  Total procedure time is determined by the timespan of the moment the patient is accepted into the room (start) and the time when the procedure is complete (finish - when physician exits room).
Accuracy of needle targeting | 24 hrs
  Distance from defined target on PercuNav and angle of entry

CONTACTS AND LOCATIONS:
Overall Officials: Edward Kim, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States